CLINICAL TRIAL: NCT07259434
Title: Time Restricted Eating in Survivors Trial 2.0
Acronym: TEST2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Amy Kirkham, Principal Investigator, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REB#47136
Record Dates: First submitted 2025-09-26; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Cardiovascular Risk; Cognitive Function; Physical Function
Keywords: Treatment; Prevention
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated to one of two groups for 16-weeks: 1) time restricted eating group + protein counselling and healthy eating education (intervention group) or 2) healthy eating education (comparison group). Participants will be randomized using an internet-based randomization service, with equal allocation to the two groups using permutated blocks with random block sizes of 2 & 4, stratified by study site, protein intake (equal to or above vs below 1.2 g/kg/day) and Framingham Risk Score (FRS; low vs moderate-high). Blinding participants to the intervention is not possible, which introduces response bias on patient-reported outcomes.
Who Masked: Outcomes Assessor
Masking Description: Individuals analyzing vascular outcome data
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time Restricted Eating (Experimental): The TRE group will be asked to restrict the time they consume food to an 8-h window starting at any time of the day and ending ≥3-h before bed, every day for 16 weeks.
  Interventions: Behavioral: Time Restricted Eating
- Healthy Eating Education (Active Comparator): The healthy eating education group will be asked not to make major changes to the timing or number of meals they consume every day for 16 weeks.
  Interventions: Behavioral: Healthy Eating Education

INTERVENTIONS:
Behavioral: Time Restricted Eating — Participants receive remote counselling on TRE and protein intake. A registered dietitian (RD) will provide counselling on protein intake to mitigate potential decreases seen with TRE. The RD will provide participants with an individualized protein intake goal and will encourage them to work toward, or maintain, consuming at least 1.2 g/kg/day. Participants will receive a reference manual with a list of foods, serving sizes and protein content to help with achieving their protein intake goal. During the intervention, participants will be asked to respond to twice-daily automated text messages with the times they started and stopped eating on that day. TRE adherence will be determined as % of days where participant responses indicate fasting for ≥16h. Protein intake adherence assessed by the RD from the 24-h diet recall. Participants will also be asked to respond with a Likert ranking (1-5) to nutrition-related texts stemming from Health Canada dietary recommendations (same as control).
  Arms: Time Restricted Eating
Behavioral: Healthy Eating Education — The initial call (week 0) will focus on healthy eating education. Each check-in call will include continued healthy eating education, collection of adverse events related to the intervention and assessment of TRE contamination (via 24-h diet recall and reporting of number and timing of meals). This information will be recorded for comparison to the TRE group and across the intervention period. To standardize the use of daily text messages and enhance study engagement, participants in the TRE and the healthy eating education groups will both be asked to respond with a Likert ranking (1-5) to a nutrition-related question stemming from the Health Canada dietary recommendations on healthy eating (e.g. "Enjoying your food is part of healthy eating. How much do you enjoy the taste of your food?" Respond with 1 to 5 where 1=do not enjoy and 5=enjoy very much).
  Arms: Healthy Eating Education

SUMMARY:
After chemotherapy, older breast cancer survivors experience a faster decline in brain function. This can make it harder to enjoy life, stay social, and maintain independence. Chemotherapy can lead to poorer lifestyle habits, like unhealthy eating, less exercise, high stress, and poor sleep. Chemotherapy can also affect important health markers like blood sugar and cholesterol. Over time, these changes can damage blood vessels, which might lead to heart and brain issues. The investigators do not fully understand why brain function declines faster after chemotherapy, especially in older survivors, because there are many factors involved. In this study, the investigators will look at how lifestyle habits (like diet, exercise, stress and sleep), health markers (like blood sugar and cholesterol), and blood vessel health (like how well blood flows and how stiff the blood vessels are) affect brain function in older breast cancer survivors. The investigators will include 152 females aged 60-85 years, who finished chemotherapy for early-stage breast cancer at least 1 year ago. The investigators will use special tests to check different parts of brain function, like language, memory, and attention, as well as brain blood vessel health. This will help to understand which factors might speed up or slow down memory and thinking problems. Since many Canadian breast cancer survivors experience faster decline in brain function after chemotherapy, this study aims to find out what might make it worse. The results could help to create better and more personalized treatment plans for older breast cancer survivors that protect brain health and reduce problems with brain function in the future.

DETAILED DESCRIPTION:
This study will be a two-centre (University of Toronto and University of Alberta), two-arm, parallel-group, randomized controlled trial in older (60+ years) breast cancer survivors.

Participants will be randomly allocated to one of two groups for 16-weeks: 1) time restricted eating group + protein counselling and healthy eating education (intervention group) or 2) healthy eating education (comparison group).

To standardize the potential participant bias toward healthy lifestyle changes and pre-existing physical activity tracking devices (i.e., Fitbits are common in this demographic), all participants will receive Canada's Food Guide, the Canadian 24-h movement guidelines, and a Garmin smartwatch at baseline. To enhance recruitment and retention, and in consideration of ethics of denying care to patients with elevated CVD risk, study staff will provide both groups with standardized healthy eating education following material from Canada's Food Guide 'Resources for Health Professionals' which aligns with dietary patterns that improve cardiovascular health. The investigators will standardize the type and frequency of intervention support across both groups but with differences in content. Support will consist of an initial call and check-in calls at weeks 1, 3, 6, 12 and daily text messages to act as a reminder, self-monitoring tool, and collect adherence. After the 16-week intervention, no further formal study support will be provided for participants. Participants will be informed they can continue to follow the interventions to the extent they choose for the next 6 months and that the investigators will contact them for one final assessment around that time. In-person study visits will include a ~4.5-h comprehensive assessment at baseline and again at 16 weeks, and one abbreviated ~2-h assessment at 40 weeks as a 24-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 60-85 years
* BMI ≥25 kg/m2
* diagnosed with early-stage (I-III) BC in the past 15 years
* received chemotherapy treatment that was completed ≥1 year earlier
* Montreal Cognitive Assessment (MoCA) score of 10-30 which aligns with no impairment to moderate impairment thresholds.

Exclusion Criteria:

* does not have a mobile device that connects to Bluetooth and can send/receive text messages
* history of physician-diagnosed heart disease, dementia or Alzheimer's disease, diabetes that requires insulin or sulfonylurea usage, or eating disorder
* MoCA total score <10 (indicating dementia)
* ≥5kg weight change within past 3 months
* taking lipid- or weight-lowering medication (e.g. statins or GLP-1 agonists)
* high-risk for malnutrition (≥3 on the Malnutrition Screening Tool)
* research MRI contraindications (e.g., pacemaker, breast tissue expander, magnetic implants)
* eating all daily calories in <10h/d in the past 3 months
* following a structured dietary practice (e.g., ketogenic diet, Weight Watchers) or actively trying to lose weight in the past 3 months
* being unable to make adjustments to eating time or nutrient intake
* regularly doing >90 min/week of moderate physical activity in the past 3 months
* severe claustrophobia
* BMI>40 kg/m2 (due to body habitus fit within MRI scanner bore)
* major psychiatric disorders (e.g. bipolar, post-traumatic stress disorder, schizophrenia)
* neurological disorders that significantly impact physical or cognitive function (epilepsy, stroke, Parkinson's disease, multiple sclerosis, amyotrophic lateral sclerosis, muscular dystrophy) or traumatic brain injury resulting in ongoing neurological deficits. If the screening process identifies patients with undiagnosed severe cognitive function (MoCA score <10) or at high risk for malnutrition (≥3 on the Malnutrition Screening Tool), the investigators will recommend that the individual see their family physician. In this process, the investigators will ask the participant if there is a family member that can also receive this information.

Ages: 60 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-10-31 (Estimated)

PRIMARY OUTCOMES:
Framingham Risk Score (10-year) | 16 weeks
  Calculated using the Canadian Cardiovascular Society's standardized scoring system where sex-specific points are assigned to age, systolic blood pressure (dependent on treatment status), HDL, total cholesterol, smoking and diabetes status. The range for females is 0-30% where a higher score indicates a greater risk of cardiovascular disease in the next 10 years.

SECONDARY OUTCOMES:
Cognitive Impairment | 16 weeks
  Assessed by Global Deficit Score (GDS). GDS is calculated as an average score from 3 tests, as described in outcomes 3, 4 and 5 below: 1) Hopkins Verbal Learning Test, 2) Trail Making Test, and 3) Controlled Oral Word Association of the Multilingual Aphasia Exam, respecitvely. Each subtest consists of a complex scoring system, detailed below, with higher values indicating greater cognitive deficits.
Cognitive Function - Verbal Learning & Memory | 16 weeks
  Assessed by the List Sorting Working Memory Test (working memory, 0-28 score range), Picture Sequence Memory Test (episodic memory, age-adjusted scale scores) and the Hopkins Verbal Learning Test (learning, memory) which includes an immediate recall, delayed recall, and recognition accuracy from a list of 12 words. Higher scores (number of correct words out of 12) are indicative of better cognitive health.
Cognitive Function - Processing Speed | 16 weeks
  Assessed by the Trail Making Test (attention, speed, executive function). Shorter test time on 2 forms of the test is indicative of better cognitive function.
Cognitive Function - Verbal Fluency | 16 weeks
  Assessed using the Controlled Oral Word Association of the Multilingual Aphasia Exam (verbal fluency). Higher total number of correct words produced within 60 seconds for each letter is indicative of better cognitive health.
Cognitive Function - Cognitive Flexibility and Attention | 16 weeks
  The Dimensional Change Card Sorting test will be used to assess individual ability to switch between tasks or rules.
Physical Function - Short Performance Battery | 16 weeks
  Participants will complete: 1) balance tests (stand for 10 sec with feet a) together, b) staggered and c) one in front of the other), 2) a chair stand test (the investigators will record how long it takes for participants to complete 5 sit to stand movements), and 3) a walking speed test (the investigators will record how long it take for participants to walk 3-4 meters at their normal walking speed). 0-12 score, with higher scores indicating higher function.
Physical Function - Six Minute Walk Test | 16 weeks
  Participants will be instructed to walk as far as possible for 6 minutes between two cones that will be placed 30-m apart. Walking distance in meters is the main outcome of the 6MWT.
Physical Function - Grip Strength | 16 weeks
  A grip strength assessment will also be administered using a dynamometer. Grip strength is commonly used in various cancer populations, including breast cancer, as a measure of upper body strength, and an indirect estimate of whole-body strength related to physical function. Dominant and non-dominant hand grip strength will be assessed as an average of 3 measurements on each side.

OTHER OUTCOMES:
Framingham Risk Score (10-year) | 6 months
  Calculated using the Canadian Cardiovascular Society's standardized scoring system where sex-specific points are assigned to age, systolic blood pressure (dependent on treatment status), HDL, total cholesterol, smoking and diabetes status. The range for females is 0-30% where a higher score indicates a greater risk of cardiovascular disease in the next 10 years.
Hemoglobin (HbA1c) | 16 weeks
  Analyzed from blood plasma using a clinical assay at a core lab
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | 16 weeks
  Calculated from fasting blood measures of glucose and insulin, analyzed using a clinical assay at a core lab.
Lipid Profile | 16 weeks, 6 months
  Total cholesterol, low-density lipoprotein (LDL), high density lipoprotein (HDL), and triglycerides analyzed from blood serum using a clinical assay at a core lab.
Liver enzymes | 16 weeks
  Alanine transaminase (ALT), aspartate aminotransferase (AST), and albumin. Analyzed from blood serum using a clinical assay at a core lab.
Brain derived neurotrophic factor (BDNF) | 16 weeks
  BDNF will be assessed via fasted venipuncture using in-house assays
Apolipoprotein E (ApoE) | 16 weeks
  ApoE will be assessed via fasted venipuncture using in-house assays
Inflammatory markers | 16 weeks
  Leptin, adiponectin, tumour necrosis factor alpha (TNF-a), Interleukin-6 (IL-6). C-reactive protein (CRP). Analyzed via fasted venipuncture using in-house assays. Markers considered together when interpreted.
Visceral Adipose Tissue (VAT) | 16 weeks
  VAT in the visceral region will be measured using 3T fat-water separation magnetic resonance imaging
Thigh Myosteatosis | 16 weeks
  Thigh muscle and intermuscular adipose tissue quantification. Measured using a custom 3T MRI sequence that provides fat-water separation and T1 maps for both thighs. Myosteatosis is calculated as fat fraction, the percent of inter and intramuscular fat in the total volume of the thigh muscle.
Thigh muscle T1 time | 16 weeks
  Measured using a custom 3T MRI sequence that provides fat-water separation and T1 maps for both thighs. T1 time will be corrected for fat and averaged over both thighs.
Liver fat fraction | 16 weeks
  Measured using a custom 3T MRI sequence that provides fat-water separation and T1 map for the 3 widest slices through the liver. Fat fraction will be calculated as the percent fat within the volume of the liver.
Liver T1 time | 16 weeks
  Measured using a custom 3T MRI sequence that provides fat-water separation and T1 map for the 3 widest slices through the liver.
Myocardium fibrosis | 16 weeks
  ECG-gated MOLLI sequence will be used for T1 mapping in a short-axis, mid-basal, left ventricular slice with T1 averaged across segments
Cerebrovascular perfusion | 16 weeks
  3D pseudo-continuous arterial spin labelling . Will be normalized to brain volume (measured via 3D T1-weighted MPRAGE sequence).
White matter hyperintensity lesion volume | 16 weeks
  Measured using T2 FLAIR sequence.
Whole brain microstructural disruptions | 16 weeks
  Measured using whole brain diffusion tensor imaging.
Hippocampus microstructural disruptions | 16 weeks
  Measured using diffusion tensor imaging for the hippocampus.
Body Composition | 16 weeks, 6 months
  Measured using a body composition device (BodPod) to estimate whole body fat (in kg and %) and fat free mass (in kg and %).
Phase Angle | 16 weeks, 6 months
  The Medical Body Composition Analyzer (mBCA;SECA mBCA 525) will be used to assess bioelectric impedance phase angle and skeletal muscle mass. Electrode stickers and wires will be placed on the participants hands and feet and bioimpedance measurements are carried out while the participant is laying down. A low alternating current will be provided, and impedance will be measured from electrode cables attached to 1) the participant's hands and feet, and 2) a measuring mat laying across the participant's knees.
Circumferences | 16 weeks, 6 months
  Waist circumference at the iliac crest will be assessed using the average of two measurements using an inelastic measuring tape. Hip circumference will be measured at the widest portion of the hips, using the average of two measurements using an inelastic measuring tape.
Blood Pressure | 16 weeks, 6 months
  Measurement of resting blood pressure 6 times, 60 seconds apart, in a standardized supine position, after 5 minutes of quiet rest. The investigators will average the 2nd through 6th measurements at each time point.
Aortic Stiffness | 16 weeks
  Aortic stiffness, measured non-invasively by pulse wave velocity, will be assessed using applanation tonometry.
Carotid Intima Media Thickness (cIMT) | 16 weeks
  Structural assessment of the carotid artery thickness will be assessed using B-mode ultrasound and artery edge-tracking software
Brachial Artery Endothelial Function | 16 weeks
  Endothelial function will be assessed using the gold standard method of flow mediated dilation (FMD) using non-invasive duplex ultrasound (GE Vivid IQ) and edge-tracking software.
Cerebrovascular Response | 16 weeks
  Cerebral blood flow velocity response (delta change compared to rest) of the middle cerebral artery will be assessed using transcranial Doppler ultrasound (Neurovision Transcranial Doppler System Model 500M) in accordance with recent guidelines, in response to postural changes (sit-to-stand) and exercise (squatting).
Physical activity tracking | through study completion, an average of 43 weeks
  A Garmin smartwatch will be used to measure Moderate-Vigorous physical activity (total minutes at each intensity), step count, sedentary time (time spent sitting).
Sleep quantity | through study completion, an average of 43 weeks
  A Garmin smartwatch will be used to measure sleep quantity (total sleep duration)
Sleep quality | through study completion, an average of 43 weeks
  A Garmin smartwatch will be used to measure sleep quality (total sleep efficiency).
Dietary Intake | 16 weeks, 6 months
  Various components of dietary intake including macronutrients and micronutrients will be assessed through 3-day food records over 2 weekdays and 1 weekend collected using ASA-24 online system
Demographics and Health History | Baseline only
  Demographics and health history questionnaire will ask participants to report their age, ethnicity, marital status, employment status, education level, house-hold income, medical history (including pregnancy complications), personal history of common comorbid conditions, family history of cardiovascular disease, smoking status (current/former/never), current medication/supplement use, exercise and rehabilitation history. Information about prior conditions and smoking, along with the blood analysis from above will be used to calculate the 10y Framingham CVD risk score.
Patient reported quality of Life | 16 weeks, 6 months
  Health-related quality of life will be patient-reported by the Medical Outcomes Study 36-item Short Form questionnaire and the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire. SF-36 scores are calculated into eight 0-100 scaled scores. Higher scores indicate better quality of life outcomes.
Fatigue | 16 weeks, 6 months
  Fatigue will be assessed by the multi-dimensional fatigue inventory (MFI) validated within cancer populations. The MFI scale is a 20-item scale. Higher total scores correspond with more acute levels of fatigue.
Sleep Quality (patient reported) | 16 weeks, 6 months
  Sleep quality will be assessed by the Pittsburgh Sleep Quality Index (19item scale), scores for each question range from 0-3, with higher scores indicating more acute sleep disturbances.
Depression and Anxiety | 16 weeks, 6 months
  Presence and severity of anxiety and depressive symptoms will be assessed using the Hospital Anxiety and Depression Scale (HADS) and the Short Form Geriatric Depression Scale (GDS). HADS consists of two subscales (0-21 for anxiety and 0-21 for depression), 0-7 indicates a normal range, 8-10 suggests the presence of, and >11 suggests probable presence of each state. GDS consists of 15 items, 0-4 is considered normal, 5-8 indicates mild depression, 9-11 indicates moderate depression, and ≥12 indicates severe depression.
Stress (subjective) | 16 weeks, 6 months
  Psychosocial stress will be measured using the Perceived Stress Scale. 10-item scale, 0-4 scoring, 0-13 is considered low stress, 14-26 is considered moderate stress, and 27-40 is considered high perceived stress.
Physical Activity (subjective) | 16 weeks, 6 months
  Physical activity habits will be assessed using the Recent Physical Activity Questionnaire (RPAQ) and the Duke Activity Status Index (DASI). RPAQ is a subjective measure of physical activity over the past four-weeks, and considered in three domains. DASI is 12-item scale, 0-58.2 scoreing, a higher score is considered a higher functional capacity.
Cognitive Impairment | 6 months
  Assessed by Global Deficit Score (GDS), which is calculated as an average of 3 tests: 1) Hopkins Verbal Learning Test, 2) Trail Making Test, and 3) Controlled Oral Word Association of the Multilingual Aphasia Exam. Each subtest consists of a complex scoring system, with higher values indicating greater cognitive deficits
Cognitive Function - Verbal Fluency | 6 months
  Assessed using the Controlled Oral Word Association of the Multilingual Aphasia Exam (verbal fluency), with higher number of words produced indicative of better cognitive health.
Cognitive Function - Verbal Learning & Memory | 6 months
  Assessed by the List Sorting Working Memory Test (working memory, 0-28 score range), Picture Sequence Memory Test (episodic memory, age-adjusted scale scores) and the Hopkins Verbal Learning Test (learning, memory) which includes an immediate recall, delayed recall, and recognition accuracy from a list of 12 words. Higher scores (number of correct words) are indicative of better cognitive health.
Cognitive Function - Processing Speed | 6 months
  Assessed by the Trail Making Test (attention, speed, executive function). Shorter test time on 2 forms of the test is indicative of better cognitive function.
Cognitive Function - Cognitive Flexibility and Attention | 6 months
  The Dimensional Change Card Sorting test will be used to assess individual ability to switch between tasks or rules.
Physical Function - Short Performance Battery | 6 months
  Participants will complete: 1) balance tests (stand for 10 sec with feet a) together, b) staggered and c) one in front of the other), 2) a chair stand test (the investigators will record how long it takes for participants to complete 5 sit to stand movements), and 3) a walking speed test (the investigators will record how long it take for participants to walk 3-4 meters at their normal walking speed). 0-12 score, with higher scores indicating higher function.
Physical Function - Six Minute Walk Test | 6 months
  Participants will be instructed to walk as far as possible for 6 minutes between two cones that will be placed 30-m apart. Walking distance in meters is the main outcome of the 6MWT.
Physical Function - Grip Strength | 6 months
  A grip strength assessment will also be administered using a dynamometer. Grip strength is commonly used in various cancer populations, including breast cancer, as a measure of upper body strength, and an indirect estimate of whole-body strength related to physical function. Dominant and non-dominant hand grip strength will be assessed as an average of 3 measurements on each side.
Height | 16-weeks, 6-months
  Measurement of height using a stadiometer, measured in metres
Body weight | 16-weeks, 6-months
  Assessed fasted in lab using a calibrated scale. Recorded in kilograms.
Body Mass Index (BMI) | 16 weeks, 6 months
  Calculated from a measurement of height and body weight to report BMI (kg/m^2)

CONTACTS AND LOCATIONS:
Overall Officials: Amy A Kirkham, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No